CLINICAL TRIAL: NCT00250263
Title: A Trial of Immunological Outcomes of Sublingual Immunotherapy for House Dust Mite (D. Pteronyssinus) Allergy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Project 170/05
Record Dates: First submitted 2005-11-06; First posted 2005-11-08 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2005-11

CONDITIONS: Allergic Rhinitis; Asthma
Keywords: rhinitis; asthma; atopy; house dust mite; immunotherapy; SLIT
MeSH Terms: conditions — Rhinitis, Allergic; Asthma; Rhinitis | interventions — Pharmaceutical Preparations; Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Placebo Comparator): Matching placebo- control arm (first year)
  Interventions: Drug: Placebo
- 2 (Active Comparator): Drug Staloral (active group)
  Interventions: Drug: (agent for immunotherapy) Staloral

INTERVENTIONS:
Drug: (agent for immunotherapy) Staloral — Immunotherapy agent for sublingual daily use. First week (vial containing the concentration 10 IR/ml) Day 1 - 1 pressure Day 2 - 2 pressures Day 3 - 4 pressures Day 4 - 6 pressures Day 5 - 8 pressures Day 6 - 10 pressures
  Second week (300 IR/ml) (vial containing the concentration 300 IR/ml) Day 7 - 1 pressure Day 8 - 2 pressures Day 9 - 4 pressures Day 10 - 6 pressures Day 11 - 8 pressures
  Maintenance phase Day 12 to 364 - 8 pressures daily
  The first year will be followed by a second year open label period (optional)- 8 pressures daily
  Arms: 2
Drug: Placebo — Matching placebo for sublingual use. Same schedule used for the intervention ACTIVE group.
  First week (vial containing placebo) Day 1 - 1 pressure Day 2 - 2 pressures Day 3 - 4 pressures Day 4 - 6 pressures Day 5 - 8 pressures Day 6 - 10 pressures
  Second week (300 IR/ml) (vial containing placebo) Day 7 - 1 pressure Day 8 - 2 pressures Day 9 - 4 pressures Day 10 - 6 pressures Day 11 - 8 pressures
  Maintenance phase Day 12 to 364 - 8 pressures daily
  Arms: 1

SUMMARY:
Allergic diseases represent a major health issue worldwide. Mainstay treatment is allergen avoidance and pharmacotherapy for symptom relief. Allergen immunotherapy offers the advantages of specific treatment with long lasting efficacy, and can modify the course of disease. However, use of this treatment is restricted by the high risk of adverse events especially in asthmatics. Other, better tolerated, routes of allergen administration than the current conventional subcutaneous route (SCIT) have been investigated including sublingual (SLIT). However, the immune parameters of SLIT have not been examined. We propose conducting a randomised, placebo-controlled study of a commercially-available SLIT for house dust mite (HDM) allergy to investigate induction of relevant T cell regulatory immune mechanisms. The first year will be followed by an optional open label extension period. Immunoregulatory cytokine synthesis and T cell phenotype and function (real time PCR and flow cytometry) will be examined. This project will provide important fundamental knowledge on which to base improved and greater application of this potentially curative treatment for allergy. SLIT has the potential advantage of home administration and suitability for patients with asthma who are currently unable to access many of the allergen desensitising regimens.

ELIGIBILITY:
Inclusion Criteria:

* allergic rhinitis and/or
* mild stable asthma
* house dust mite allergic
* positive HDM-specific IgE as determined by skin prick test (wheal diameter >6 mm to D. pteronyssinus) or CAP-Pharmacia score > 2

Exclusion Criteria:

* Immunodeficiency diseases
* Severe or uncontrolled asthma
* Previous immunotherapy with House dust mite (HDM) extract within the last five years or ongoing immunotherapy with HDM or other allergens
* Continuous oral corticosteroids
* Subjects on treatment with beta-blockers
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Immunological mechanisms of SLIT by phenotyping different subsets of cytokine positive T cells, regulatory T cells, and memory T cells in peripheral blood of subjects before, during and after immunotherapy. | 12 and 24 months
-Expression of "immunoregulatory" cytokines by CD4+ T | 12 and 24 months
cells | 12 and 24 months
- Helper, regulatory and memory T cell subsets | 12 and 24 months
(a) Helper T cells | 12 and 24 months
(b) Regulatory T cells | 12 and 24 months
b1- Regulatory T cell phenotype | 12 and 24 months
b2- Regulatory T cell function | 12 and 24 months

SECONDARY OUTCOMES:
Symptom diary, medication use, visual analogue score, disease-specific rhinoconjunctivitis Quality of Life Questionnaire | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Robyn O'Hehir, MD FRACP FRCP PhD, Principal Investigator — Alfred Hospital; Monash University; Jennifer Rolland, PhD, Study Chair — Alfred Hospital; Monash University; Jo Douglass, MBBS FRACP MD, Study Chair — Alfred Hospital; Monash University
Locations (1):
- The Alfred Hospital. Department of Allergy Immunology & Respiratory Medicine, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Fanta C, Bohle B, Hirt W, Siemann U, Horak F, Kraft D, Ebner H, Ebner C. Systemic immunological changes induced by administration of grass pollen allergens via the oral mucosa during sublingual immunotherapy. Int Arch Allergy Immunol. 1999 Nov;120(3):218-24. doi: 10.1159/000024270. PMID 10592467
- [Background] Gardner LM, Thien FC, Douglass JA, Rolland JM, O'Hehir RE. Induction of T 'regulatory' cells by standardized house dust mite immunotherapy: an increase in CD4+ CD25+ interleukin-10+ T cells expressing peripheral tissue trafficking markers. Clin Exp Allergy. 2004 Aug;34(8):1209-19. doi: 10.1111/j.1365-2222.2004.02009.x. PMID 15298560
- [Background] Rolland JM, Douglass J, O'Hehir RE. Allergen immunotherapy: current and new therapeutic strategies. Expert Opin Investig Drugs. 2000 Mar;9(3):515-27. doi: 10.1517/13543784.9.3.515. PMID 11060692
- [Derived] O'Hehir RE, Gardner LM, de Leon MP, Hales BJ, Biondo M, Douglass JA, Rolland JM, Sandrini A. House dust mite sublingual immunotherapy: the role for transforming growth factor-beta and functional regulatory T cells. Am J Respir Crit Care Med. 2009 Nov 15;180(10):936-47. doi: 10.1164/rccm.200905-0686OC. Epub 2009 Aug 20. PMID 19696440